CLINICAL TRIAL: NCT02629081
Title: Image-Enhanced Endoscopy for the Diagnosis of Non-Erosive Reflux Disease: A Prospective Case-Control Trial
Brief Title: Image-Enhanced Endoscopy (IEE) for Diagnosis of Non-Erosive Reflux Disease
Status: Completed | Type: Observational
Sponsor: Loren Laine (Other)
Responsible Party: Sponsor-Investigator, Loren Laine, Professor of Medicine, Digestive Diseases, Yale University
Organization: Yale University (Other)
Other Study IDs: HIC1503015486; 0005 (Other: VACHS)
Record Dates: First submitted 2015-12-08; First posted 2015-12-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: GERD
Keywords: heartburn; GERD; NERD; non-erosive reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Non-Erosive Reflux Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Controls & Cases: Controls (participants without heartburn or other GERD symptoms undergoing standard upper endoscopy for the following: anemia, weight loss, diarrhea, and screening for esophageal varices) and Cases (participants with heartburn or other GERD symptoms undergoing standard endoscopy for heartburn or other GERD symptoms.)
  Interventions: Other: Controls & Cases

INTERVENTIONS:
Other: Controls & Cases — All interventions are standard of care and both controls and cases will be treated the same. IEE results from controls and cases will be compared.

SUMMARY:
When treating persistent heartburn from gastroesophageal reflux disease (GERD) that does not respond to conventional treatment (a class of medications called proton pump inhibitors), it is important to be able to distinguish between erosive GERD and non-erosive GERD (called NERD).

Currently the best method the investigators have to make this distinction is esophageal 24-hour pH and impedance testing. The test involves inserting a catheter into the esophagus through the nose and having the catheter maintained in this position for 24 hours This test is invasive, can be uncomfortable, and it is expensive and time consuming.

The investigators are hoping that image enhanced technology will identify characteristics that are found more commonly in patients with non-erosive GERD compared to controls and therefore provide evidence that may allow us to replace pH and impedance testing with the image enhanced endoscopy as the best way to diagnose NERD.

Participants will be either patients undergoing an upper endoscopy as part of their standard clinical evaluation for heartburn that does not respond to PPIs or patients undergoing standard clinical evaluation endoscopy for other reasons.

DETAILED DESCRIPTION:
Evaluation of the utility of image-enhanced endoscopy (IEE) in the diagnosis of non-erosive reflux disease (NERD), defined as heartburn documented to be associated with reflux on impedance-pH testing in the absence of erosions on standard white-light endoscopy (WLE) during initial endoscopy.

The investigators will examine the following characteristics for IEE sensitivity, specificity, positive predictive values, and negative predictive value: squamo-columnar junction (SCJ) vascularity, micro-erosions, SCJ pit pattern, and combinations of these characteristics. The investigators will also look at abnormal morphology of intra-papillary capillary loops (IPCLS) using the newer generation Narrow Band Light (NBI-190 endoscopes and assess the identification of their presence using I-scan. Additionally, the investigators will examine real-time diagnostic yield of reflux diseases by IEE (in vivo diagnosis of reflux disease) and analyze obtained images and results to calculate inter-observer agreement.

IEE utilized will be commonly available I-scan (Pentax) and Narrow Band Imaging (Olympus).

Consecutive patients who meet eligibility criteria and are scheduled for upper endoscopy at locations specified in this record will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an upper endoscopy for anemia, weight loss, diarrhea, or screening for esophageal varices without heartburn or other GERD symptoms and patients scheduled for upper endoscopy for heartburn not resolving with PPIs

Exclusion Criteria:

* Patients who have evidence of erosive esophagitis under white-light endoscopy
* Patients with Barrett's esophagus or esophageal malignancy on prior or current endoscopy
* Patients unable or unwilling to sign informed consent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Controls (participants scheduled for upper endoscopy for anemia, weight loss, diarrhea, or screening for esophageal varices and who do not have heartburn or other GERD symptoms and Cases (participants scheduled for upper endoscopy for heartburn or other GERD symptoms.)
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Squamo-columnar junction vascularity (graded as present or absent by endoscopist using IEE) | Once--at endoscopy

SECONDARY OUTCOMES:
Presence or absence of micro-erosions identified by endoscopist using IEE | Once at endoscopy
Squamo-columnar junction pit pattern (graded as round or non-round by endoscopist using IEE) | Once at endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Loren Laine, MD, Principal Investigator — Yale University, VACHS
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - VACHS, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Undecided